CLINICAL TRIAL: NCT02471859
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending, Single- and Multiple-Oral-Dose, Safety, Tolerability, and Pharmacokinetic Study of GDC-3280 in Healthy Subjects
Brief Title: A Safety, Tolerability, and Pharmacokinetic Study of GDC-3280 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GB29751; 2015-000560-33 (EudraCT Number)
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Part A: GDC-3280 (Experimental): Participants in multiple cohorts and treatment periods will receive single doses of GDC-3280 under fed/fasting conditions.
  Interventions: Drug: GDC-3280
- Part A: Placebo (Placebo Comparator): Participants in multiple cohorts and treatment periods will receive single doses of placebo under fed/fasting conditions.
  Interventions: Drug: Placebo
- Part B: GCD-3280 (Experimental): Participants in different cohorts will receive GDC-3280 in multiple ascending doses under fed/fasting conditions.\n
  Interventions: Drug: GDC-3280
- Part B: Placebo (Placebo Comparator): Participants in different cohorts will receive placebo in multiple ascending doses under fed/fasting conditions.\n
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GDC-3280 — GDC-3280 at various doses, depending on the cohort and treatment period
  Arms: Part A: GDC-3280; Part B: GCD-3280
Drug: Placebo — Placebo at various doses, depending on the cohort and treatment period
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
This is a Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending, Single- and Multiple-Oral Dose, Safety, Tolerability, and Pharmacokinetic Study of GDC-3280 in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female, using highly effective contraception
* Has a body mass index (BMI) 18.0 to 30.0 kg/m2, inclusive
* Is in good general health
* Having signed informed consent, is willing and able to comply with requirements of the study

Exclusion Criteria:

* Does not satisfy all screening criteria per protocol
* Is employed by or related to any personnel involved in the trial
* Has any history or condition that per protocol or in the opinion of the investigator could compromise the participant's safety or analysis of results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing an adverse event | Up to approximately 6 months

SECONDARY OUTCOMES:
Maximum concentration (Cmax) for GDC-3280 | Up to 4 days
Time to Cmax (Tmax) for GDC-3280 | Up to 4 days
Total serum clearance for GDC-3280 | Up to 4 days
Volume of distribution for GDC-3280 | Up to 4 days
Elimination half-life for GDC-3280 | Up to 4 days
Serum GDC-3280 concentration-time data by dosing group | Up to 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Leeds, United Kingdom